CLINICAL TRIAL: NCT01144754
Title: A Prospective Observational Study of Newly Diagnosed Diffuse Large B Cell Primary Breast Lymphomas Treated With RCHOP With or Without Radiotherapy
Brief Title: Observational Study of Diffuse Large B Cell Primary Breast Lymphomas Treated With RCHOP +/- XRT
Status: Terminated | Type: Observational
Why Stopped: Low Accrual
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: LYMNHL0071; SU-03042009-1939 (Other: Stanford University)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — Calculated per patient
  Other Names: Rituxan; MabThera

SUMMARY:
This is a multi-center observational study to assess addition of Rituximab in the treatment of previously untreated patients with Diffuse Large B-Cell Lymphomas(DLBCL) over an enrollment period of 60 months. Patients in this study are enrolling for the collection of their data on observations made during normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with DLBCL of the breast.
* Patients must have CD20 positive tumors.
* Stage IE or IIE.
* Must have at least one objective measurable or evaluable disease. Baseline measurements and evaluations must be obtained within 4 weeks of registration to the study.
* Patients must not have historical or radiographic evidence of CNS metastasis including previously treated, resected or asymptomatic brain lesions or leptomeningeal involvement.
* Patients must have an ECOG performance status 0-2.
* Patients must have adequate organ function as evidenced by the following laboratory studies (within 2 weeks prior to registration):

  * Creatinine Clearance >= 50 ml/min
  * Total bilirubin <= 2.0 mg/dl and AST <= 2 x upper limit of normal. If documented hepatic involvement with lymphoma, total bilirubin can be <= 3 x *ULN, and AST <= 5 x ULN.
  * Absolute neutrophil count >= 1500/mm3 and platelet count >= 100,000/mm3. If documented bone marrow involvement with lymphoma, absolute neutrophil count >= 500/mm^3 and platelet count >= 50,000/mm^3.
* Patients must be age >= 18 years.
* Women must not be pregnant or breast feeding due to potential harmful effects to the fetus/baby. Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception.
* Patients must not have an active infection requiring parental antibiotics.
* Patients with known HIV infection are excluded.
* Patients must have a normal left ventricular ejection fraction to be eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated patients with DLBCL of the breast.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N. Ganjoo, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States